CLINICAL TRIAL: NCT01637571
Title: The Effect of Dexilant Treatment on Esophageal Hypersensitivity in GERD Related Non Cardiac Chest Pain Patients
Brief Title: Dexilant Treatment in Gastrointestinal Reflux Disease (GERD Related Non Cardiac Chest Pain
Acronym: Dexilant
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor could not fund
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201102718
Record Dates: First submitted 2011-12-06; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Chest Pain; Gastrointestinal Reflux Disease
Keywords: GERD; NCCP; chest pain; reflux; GERD related non-cardiac chest pain
MeSH Terms: conditions — Chest Pain; Gastroesophageal Reflux | interventions — Dexlansoprazole

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Dexilant (Active Comparator): 60mg of Dexilant QD for 12 weeks
  Interventions: Drug: Dexilant
- Placebo (Placebo Comparator): 60mg of Dexilant placebo QD for 12 weeks
  Interventions: Drug: Dexilant Placebo

INTERVENTIONS:
Drug: Dexilant — 60mg of Dexilant QD for 12 weeks
  Arms: Dexilant
Drug: Dexilant Placebo — 60mg of Dexilant placebo QD for 12 weeks
  Other Names: Dexlansoprazole
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate a new treatment for non-cardiac chest pain (NCCP) related to gastrointestinal reflux disease (GERD), called Dexilant. The investigators would like to test its effectiveness in treating NCCP.

The patient will undergo esophageal balloon distention testing (EBDT) before and after taking the new treatment for one month (Dexilant). EBDT evaluates the sensation and mechanical properties of the esophagus. A catheter with a deflated balloon is placed through the mouth and into the esophagus and the balloon is inflated with water. ECG and labs will be done throughout the study as a measurement of safety.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years
2. NERD, or GERD LA Class A-B (endoscopy)
3. Subjects with positive pH testing
4. At least one episode of chest pain a week in the past month
5. Previous negative cardiac evaluation (EKG ± stress test ± coronary angiogram)
6. Negative esophageal evaluation for a motility disorder (Nutcracker esophagus, achalasia)

Exclusion Criteria:

1. Subjects requiring narcotics or other pain medications, Subjects with known LA class C-D, Barrett's esophagus or peptic stricture on endoscopy
2. Subjects with previous upper gastrointestinal surgery
3. Pregnancy
4. Subjects with diabetes, neuromuscular disorders, or other severe co-morbidities
5. (Cardiovascular, respiratory, renal, hepatic, hematologic, endocrine, neurologic, and psychiatric).
6. Subjects with upper airway symptoms (such as hoarseness, wheezing, laryngospasm).
7. Medications such as baclofen, and prokinetic agents.
8. History of substance abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Frequency of chest pain episodes in treatment vs placebo groups | 12 weeks
  the number of chest pain episodes during the study

SECONDARY OUTCOMES:
Intensity of chest pain episodes | 12 weeks
  how strong the chest pain episodes are
Sensory thresholds for first sensation | 12 weeks
  the balloon distension level when a sensation is first felt
Sensory thresholds for discomfort | 12 weeks
  the balloon distension level when discomfort is felt
Sensory thresholds for pain | 12 weeks
  the balloon distension level when pain is felt
duration of chest pain episodes | 12 weeks
  how long the chest pain episodes last

CONTACTS AND LOCATIONS:
Overall Officials: Ron Schey, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States